CLINICAL TRIAL: NCT06168006
Title: Effects of a Physical Training Program Using a Mobile App on the Functionality and Cardiovascular Function of Individuals With Post-covid-19 Syndrome: Randomized Clinical Trial
Brief Title: Exercise Training Using an App on Physical Cardiovascular Function Individuals With Post-covid-19 Syndrome
Acronym: Recovery
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nove de Julho (Other)
Responsible Party: Principal Investigator, Raphael Mendes Ritti Dias, Professor, University of Nove de Julho
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Recovery Long Covid
Record Dates: First submitted 2023-12-12; First posted 2023-12-13 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Post-Acute COVID-19 Syndrome
Keywords: exercise; mobile app; physical function; cardiovascular function
MeSH Terms: conditions — Post-Acute COVID-19 Syndrome; Motor Activity | interventions — Exercise; Rehabilitation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Outcomes assessor will be blinded for the group of the subjects
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise intervention (Experimental): The subjects randomized to this group will perform three app-based training sessions per week for 12 weeks, each session lasting a maximum of 40 minutes.
  Interventions: Behavioral: Exercise
- Control intervention (Sham Comparator): This group will receive a booklet with exercise instructions, and will be recommended the same frequency and duration of exercise as the experimental group
  Interventions: Behavioral: Control

INTERVENTIONS:
Behavioral: Exercise — The experimental group will undergo an exercise program using the Recovery App. Participants will receive guidance from researchers about the functionality of the app. The Recovery App includes flexibility, strength, and aerobic training exercises, aiming for a progressive intensity and volume over the weeks.
  Other Names: Rehabilitation; Physical activity; Endurance; Resistance exercises
  Arms: Exercise intervention
Behavioral: Control — They will receive an exercise booklet based on the Brazilian Physical Activity Recommendations (MINISTRY OF HEALTH, 2021), which recommend 150 minutes of physical activity for adults and seniors.
  Arms: Control intervention

SUMMARY:
The aim of this study is to assess the effect of a physical exercise program via a mobile application on functional parameters in individuals with post-COVID-19 syndrome. This is a clinical trial involving 60 individuals with post-COVID syndrome who will be randomly assigned to either a control group (physical activity guideline) or an experimental group (app-based training).

ELIGIBILITY:
Inclusion Criteria:

* Laboratory diagnosis of COVID-19
* Fatigue ≥ 8 points on the Chalder Scale and/or dyspnea 2-4 on the Modified Medical Research Council
* Have access to a smartphone
* Have no contraindications for exercise practice
* Have ability to sit and stand and maintain balance while standing
* Have preserved cognitive function
* Have no risk of falls according to the Morse Fall Scale

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-03-01 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in 6 min-walk test distance at 12 weeks | Baseline and 12 weeks
  The 6-minute walk test performed in a 30-meter corridor, measured in meters
Change from baseline in Glittre test at 12 weeks | Baseline and 12 weeks
  The test consists in rise from a chair, carry a weighted backpack, walk 10 meters, climb stairs, move objects between shelves (1 kg each), and return. They perform tasks sequentially, transferring items up and down shelves. The route is retraced, ending by sitting back in the initial chair, measured in seconds
Change from baseline in sit and stand test at 12 weeks | Baseline and 12 weeks
  The test consists in rising from a chair as many times as possible within 30 seconds, measured in number of repetitions
Change from baseline in Post-Covid Functional Scale at 12 weeks | Baseline and 12 weeks
  The Post-COVID-19 Functional Status Scale assesses limitations following SARS-CoV-2 infection, measured as a score

SECONDARY OUTCOMES:
Change from baseline in Patient Functional Scale at 12 weeks | Baseline and 12 weeks
  The Patient Functional Scale allows individuals to identify 3 to 5 important activities they consider themselves unable to perform or are having difficulty with due to their condition, measured in a score
Change from baseline in Motor Evoked Potential at 12 weeks | Baseline and 12 weeks
  The cortical excitability of the quadriceps motor area will be measured using Motor Evoked Potential results in microvolts (µV) using the Transcranial Magnetic Stimulation equipment model MagPro R20 (MagVenture, Denmark) with the parabolic coil model MMC-140-II, measured in kgf
Change from baseline in Modified Medical Research Dyspnea Scale at 12 weeks | Baseline and 12 weeks
  This scale comprises five items, allowing the patient to select the item that corresponds to how much their dyspnea limits their daily life activities, measured as a score
Change from baseline in Chalder Physical Fatigue Scale at 12 weeks | Baseline and 12 weeks
  Comprising eight specific statements about physical fatigue to confirm its presence or absence, measured as a score
Change from baseline in De Paul Symptom Questionnaire at 12 weeks | Baseline and 12 weeks
  The questionnaire evaluate the symptoms of fatigue in different conditions, measured as a score
Change from baseline in Quality of Life at 12 weeks | Baseline and 12 weeks
  To assess quality of life, the 12-Item Short-Form Health Survey will be used, consisting of twelve items that evaluate eight different dimensions influencing quality of life, measured as a score
Change from baseline in Frailty and Sarcopenia at 12 weeks | Baseline and 12 weeks
  Frailty will be assessed using the Tilburg Frailty Indicator, while sarcopenia will be evaluated through the Sarcopenia Form questionnaire, both measured as a score
Change from baseline in Anxiety and Depressive Symptoms at 12 weeks | Baseline and 12 weeks
  Levels of anxiety and depression will be assessed using the Hospital Anxiety and Depression Scale, measured as a score
Change from baseline in Pain at 12 weeks | Baseline and 12 weeks
  Assessed using the Numeric Pain Rating Scale, measured as a score
Change from baseline in Movement Behavior at 12 weeks | Baseline and 12 weeks
  Movement behavior will be quantified through a motion sensor, measured in minutes
Change from baseline in Barriers to Physical activity at 12 weeks | Baseline and 12 weeks
  Specific questionnaire to assess the most prevalent environmental barriers to physical activity, measured as presence or absence
Post assessment of Exercise Adherence Assessment Scale | 12 weeks
  Adherence to exercise interventions will be obtained with the Adherence Assessment Scale
Change from baseline in Blood Pressure at 12 weeks | Baseline and 12 weeks
  The clinical resting blood pressure will be assessed using automatic blood pressure monitoring equipment (HEM-7113, OMRON®, Brazil), measured in mmHg
Change from baseline in Cardiac Autonomic Modulation at 12 weeks | Baseline and 12 weeks
  Cardiac autonomic modulation will be assessed through heart rate variability using a heart rate monitor, measured in RR intervals
Change from baseline in Blood Flow and Flow-mediated Dilation at 12 weeks | Baseline and 12 weeks
  The measurements of basal blood flow and flow-mediated vasodilation will be obtained through ultrasonography in brachial artery, measured in ml/min or %
Change in Spirometry parameters at 12 weeks | Baseline and 12 weeks
  Changes in Forced vital capacity, forced expiratory volume in the first second, Peak expiratory flow, forced expiratory flow 25-75% and FEV 1 /FVC ratio

OTHER OUTCOMES:
System Usability Scale | 12 weeks
  Scale used to assess the individuals' perception of the app's usability in the group submitted to the intervention
The User Experience Questionnaire | 12 weeks
  The questionnaire will be applied in experimental group to collect information regarding the user's overall experience with the app, such as: general perception, overall experience, main barriers, and key difficulties in using the app.
Focal group | 12 weeks
  The focus group will be conducted via video conference with 4 to 10 individuals that participated in experimental group. The guiding questions will aim to understand the user's perception, from usability to effectiveness, including satisfaction and potential improvements to the app.

CONTACTS AND LOCATIONS:
Overall Officials: Fernanda Corrêa, PhD, Principal Investigator — University of Nove de Julho
Locations (1):
- Universidade Nove de Julho, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Yes
The data will be available after the completion of the study and the finalization of the main articles of this projects
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: After the publication of the main articles of the study.
Access Criteria: Upon reasonable request